CLINICAL TRIAL: NCT07283497
Title: Itraconazole Therapy In Bronchiectasis With Airway Mold: A Single-Arm Pilot Trial Of Feasibility, Safety, And Impact On Respiratory Symptoms And Airway Microbiome Diversity
Brief Title: Itraconazole Therapy In Bronchiectasis With Airway Mold
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amjad Kanj, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-010613
Record Dates: First submitted 2025-12-01; First posted 2025-12-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Bronchiectasis; Fungal Infection of Upper Respiratory Tract
MeSH Terms: conditions — Bronchiectasis | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bronchiectasis (Experimental): Subjects with bronchiectasis and airway mold
  Interventions: Drug: Itraconazole 200 mg

INTERVENTIONS:
Drug: Itraconazole 200 mg — Subjects will receive oral itraconazole, 200 mg twice daily, for six weeks, based on prior dosing regimens for airway fungal disease.

SUMMARY:
The primary objective of this study is to evaluate the feasibility of itraconazole therapy in patients with bronchiectasis and airway mold. Feasibility will be assessed through recruitment success, treatment adherence, tolerability, and participant retention. The study will also explore the impact on respiratory symptoms and airway microbiome diversity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years seen at Mycobacterial and Bronchiectasis Clinic (MMBC) in Rochester
* Diagnosis of bronchiectasis confirmed by MMBC provider and chest CT
* Within the last 3 months - culture growth of a mold in high quantity ('many') or culture growth of at least two distinct mold species in any quantity
* Not actively on antimicrobial therapy AND no current plan to initiate antimicrobial therapy at the time of enrollment, as determined by treating provider
* Ability to produce spontaneous sputum at Visit 1.

Exclusion Criteria:

* Known diagnosis of allergic bronchopulmonary aspergillosis or invasive fungal disease
* Use of the following medications: rifampin, rifabutin, phenobarbital, phenytoin, carbamazepine, dofetilide, quinidine, dronedarone, simvastatin, lovastatin, certain immunosuppressants (tacrolimus, cyclosporine, sirolimus, everolimus) and anticoagulants (rivaroxaban, apixaban, edoxaban, warfarin).
* Abnormal baseline liver function tests (ALT, AST, alkaline phosphatase, or bilirubin > upper limit of normal)
* Prolonged QTc interval on baseline ECG (>460 ms in females or >450 ms in males)
* History of congestive heart failure (black box warning), known cardiomyopathy, or arrhythmias
* Pregnancy or lactation
* Known hypersensitivity or contraindication to azole antifungal therapy
* Prior use of systemic antifungals within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible patients who consent and enroll | 2 years
  Recruitment will be measured as the proportion of eligible patients who consent and enroll out of patients screened, reported as a percentage, with a benchmark of >60%.
Number of patients to achieve successful medication adherence | 2 years
  Adherence will be assessed through pill counts with successful adherence defined as ≥ 70% of doses taken and achieving a therapeutic trough level.
Proportion of participants who complete treatment without adverse effects | 2 years
  Tolerability will be evaluated as the proportion of participants who complete the 6-week course without discontinuation due to adverse effects, with a target benchmark of ≥ 70%.
Proportion of patients retained for complete study | 2 years
  Retention will be defined as the proportion of participants completing all scheduled study visits (baseline, day 7 and end of treatment), with a goal of ≥ 80% retention.

SECONDARY OUTCOMES:
Number of participants meeting hepatic safety discontinuation criteria | Baseline, 1 week
  Hepatic safety will be monitored with serial hepatic function panels obtained at baseline, day 7, with the endpoint defined as the number of participants meeting discontinuation criteria: total bilirubin more than 2 times the ULN according to Mayo laboratory reference, ALT more than two times the ULN, AST more than two times the ULN, or ALP greater than 250 U/L.
Number of participants with a QTc interval greater than 500 ms | Baseline, 1 week
  Cardiac safety will be assessed by obtaining an ECG on day 7, with the endpoint defined as the proportion of participants with a QTc interval greater than 500 ms.

CONTACTS AND LOCATIONS:
Overall Officials: Amjad Kanj, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials